CLINICAL TRIAL: NCT06101238
Title: BLOODSAFE- Implementation of Iron Supplementation and Nutritional Counselling Interventions to Improve Availability and Safety of Blood in Ghana-a Type I Pragmatic Effectiveness- Implementation Hybrid Trial
Brief Title: BLOODSAFE Ghana- Iron and Nutritional Counselling Strategy
Acronym: UH3BLIS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: University of Ghana (Other); National Blood Service Ghana (Other); Syracuse University (Other); Liverpool School of Tropical Medicine (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: B08; UH3HL151599-04 (NIH)
Record Dates: First submitted 2023-10-11; First posted 2023-10-26 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Blood Donation
MeSH Terms: interventions — Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Iron Supplementation (Experimental)
  Interventions: Dietary Supplement: supplementation with low dose elemental iron
- Standard of Care (No Intervention)

INTERVENTIONS:
Dietary Supplement: supplementation with low dose elemental iron — 65mg daily
  Arms: Iron Supplementation

SUMMARY:
A randomized trial will compare 6-months of low-dose (65mg elemental iron daily) among prospective blood donors who are deferred for low haemoglobin but have passed all of the other pre-screening requirements for blood donation to a group of donors who were deferred from donating and receive the current standard of care (nutrition counseling only). An automated full blood count (FBC) will also be done to identify any safety concerns. The randomized trial will evaluate effectiveness with the primary outcome of at least one successful donation during a 12-month follow-up period. Safety will be evaluated by tracking iron supplementation related adverse events (e.g., lower gastrointestinal) and acceptability (e.g., compliance to study prescribed regimen) with monthly phone calls. Participants will be followed for a total of 12 months from screening with follow up phone calls at 4 weekly intervals. All participants will receive nutrition counselling and haemoglobin will be evaluated at screening. Individuals with very low haemoglobin (<10g/dl in females and <11g/dl in males) will be identified by an automated FBC at screening and referred for proper medical care.

Sample size will be 264 per group: this gives 80% power for detecting an odds ratio of 2.6. With 2 donors recruited at each donation event, this will require 264 donation events. This corresponds to 2.5 donation events per week for 2 years or 2 donation events per week for 2.5 years.

ELIGIBILITY:
Inclusion Criteria:

* individuals between 18 - 60 years who weigh at least 50kg
* pass pre-donation screening using the NBSG standardized donor screening questionnaire
* vital signs meet the NBSG requirement for blood donation
* non-contact forehead temperature not exceeding 37.5°C
* meeting acceptable requirements for skin lesions, needle marks and physical appearance.
* willingness and ability to consent
* understands one of English, Twi, Ewe, or Ga
* deferred for low haemoglobin
* intend to remain in the study during the entire length of the study

Exclusion Criteria:

* persons who have used iron supplementation within the past one month
* potential donors who are found to have haemoglobin Hb < 10g/dl (females) and Hb<11g/dl (males) at screening

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 533 (Actual)
Dates: Start 2024-01-11 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with a successful blood donation | 12 months

SECONDARY OUTCOMES:
Proportion of participants who attempt blood donation | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
The BLOODSAFE project is committed to quickly sharing results and data. Papers will be submitted summarizing the primary results of the BLOODSAFE studies once the analysis is complete. These results will be published in major scientific journals and presented at scientific meetings.